CLINICAL TRIAL: NCT04473937
Title: Radiation Therapy To Enhance CAR T Efficacy Early in Post-CAR T Cell Therapy Refractory Lymphoma: A Pilot Study
Brief Title: Radiation Post-CAR T in Refractory Lymphoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Chirayu Patel, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-861
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Malignancy; Refractory Lymphoma
Keywords: Hematologic Malignancy; Refractory Lymphoma; CAR T cell therapy; Radiotherapy
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Radiotherapy (Experimental): Participants must have received CAR-T infusion within the last 90 days prior to completing a study screening and enrollment process.
  * Participants will be enrolled within 28 days after screening is complete and radiotherapy will occur within 14 days after study enrollment.
  * Radiotherapy will be administered based on a dose and schedule pre-determined by the study doctor.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy at pre-determined dose and schedule

SUMMARY:
This study is evaluating the safety and efficacy of using radiotherapy in participants who have refractory lymphoma shortly after receiving CAR T cell therapy (axicel or tisacel).

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this intervention after administration of CAR T cell therapy. This research study looks to systematically investigate the safety and efficacy of radiotherapy following CAR T cell therapy (axicel or tisacel) in refractory lymphoma. CAR T cell therapy involves genetically modifying T cells to target tumor cells for death. Radiotherapy is a standard treatment offered with refractory lymphoma and uses high-energy x rays, or particles, to destroy or damage cancer cells. Few have received CAR T cell therapy prior to radiation therapy and this study aims to gather more information on radiotherapy following CAR T cell therapy as a treatment option and its potential to improve participants immune system's response to cancer cells as well as its interaction with CAR T cell therapy to better treat refractory lymphoma.

The research study procedures include screening for eligibility, enrollment, biopsy following radiation, post-treatment period, and long-term follow-up.

* Participants will receive radiotherapy at a dose and schedule determined by the study doctor.
* Participants will be followed for up to 24 months after completion of study treatment.

It is expected that about 20 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to undergo biopsy. Biopsy will be obtained for patients to exclude possibility of false negative residual FDG avidity on PET/CT that is not substantially increased relative to pre-CAR-T PET/CT. Exceptions are allowed for patients who have clearly progressive disease for whom delaying radiation therapy to obtain a biopsy may worsen outcome (such as cases of cord compression), and for patients for whom the risks of biopsy are high (such as patients with evidence for CNS involvement).
* Biopsy-confirmed refractory disease within 30-90 days following commercial axicabtagene ciloleucel or tisagenlecleucel therapy for a hematologic malignancy (these include relapsed or refractory large B-cell lymphoma after two or more lines of systemic therapy, including diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma, and DLBCL arising from follicular lymphoma). Of note, 'refractory' refers to patients who had early refractory disease after CAR-T cell therapy and not to patients who have received CAR-T for refractory disease, but had complete response to CAR-T cell therapy.
* At least 1 measurable lesion according to the Lugano criteria1. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy
* The following criteria pertain to pattern of progression:

  * Patients may have one refractory lesion without other residual or progressive disease as per PET/CT
  * Patients may have more than one refractory lesion, but with evidence for at least partial response of at least one other lesion as per PET/CT
  * Patients with more than one site of refractory disease without evidence for at least partial response of at least one other lesion are eligible if they are:

    * A. Symptomatic from a refractory lesion (such as cord compression or focal pain) or
    * B. Have disease that can locally affect the spinal canal or brain if left untreated.
* Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for clinically non-significant toxicities such as alopecia and prolonged cytopenias that are not expected to worsen during RT) if there is concern for overlap of anticipated radiation-related toxicity and toxicity from prior therapy due to where the RT field is located.
* Age 18 or older
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Any medical condition likely to interfere with assessment of safety or efficacy of RT
* Patients with more than one site of disease without any evidence for response to CAR T cell therapy who are not focally symptomatic due to progressive disease or do not have disease that can locally affect the spinal canal or brain if left untreated
* Women of child-bearing potential who are pregnant because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential.
* In the investigators judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-10-09 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chirayu G Patel, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiotherapy: Participants must have received CAR-T infusion within the last 90 days prior to completing a study screening and enrollment process.
  * Participants will be enrolled within 28 days after screening is complete and radiotherapy will occur within 14 days after study enrollment.
  * Radiotherapy will be administered based on a dose and schedule pre-determined by the study doctor.
  Radiotherapy: Radiotherapy at pre-determined dose and schedule
Period: Overall Study
Arm/Group | Radiotherapy
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiotherapy
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 79 [78 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2
  Hispanic | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0
Description: Rate and severity of radiotherapy-related toxicity as per CTCAE v5.0 (Common Terminology Criteria for Adverse Events) during radiotherapy (RT) or within the first 30 days of completing RT. The number of participants who experienced radiotherapy-related toxicities are listed below.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy
Number analyzed (Participants) | 3
Participants
  Grade 2 dermatitis | 1
  Grade 1 Dysgeusia | 1
  Grade 1 Skin hyperpigmentation | 1
  Grade 1 Skin ulceration | 1
  Grade 1 Anorexia | 1
  Grade 1 Neck Edema | 1
  Grade 1 Fatigue | 1
  Grade 1 Nausea | 1
  Total number of participants who experienced one or more RT-related toxicities, as described above | 2

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the length of time between a subject's first objective response per Lugano criteria (complete response or partial response) and local disease progression per Lugano criteria, or death regardless of cause.
Time Frame: Up to 2 years
Measure: Mean (Full Range); unit: months
Arm/Group | Radiotherapy
Number analyzed (Participants) | 3
months | 7.33 [0 to 22]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the incidence of either a complete response or a partial response by Lugano criteria. All subjects that do not meet the criteria for an objective response by the analysis data cutoff date will be considered non-responders.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy
Number analyzed (Participants) | 3
Participants | 3

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from radiotherapy completion date to the date of disease progression per Lugano criteria or death from any cause. Subjects not meeting the criteria for progression by the analysis data cutoff date will be censored at their last evaluable disease assessment date.
Time Frame: Up to 2 years
Measure: Mean (Full Range); unit: months
Arm/Group | Radiotherapy
Number analyzed (Participants) | 3
months | 0.67 [0 to 2]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from radiotherapy completion to the date of death. Subjects who have not died by the analysis cutoff date will be censored at their last contact date.
Time Frame: Up to 2 years
Measure: Mean (Full Range); unit: months
Arm/Group | Radiotherapy
Number analyzed (Participants) | 3
months | 7.33 [0 to 22]

ADVERSE EVENTS:
Time Frame: All adverse events are reported from enrollment through 3 months after radiation therapy. After 3 months, targeted adverse events (neurological, hematological, infections, autoimmune disorders, and secondary malignancies) are reported for 6 months after treatment with axicel or tisacel or until disease progression, whichever occurs first. All cause mortality was monitored for up to two years.
Arm/Group | Radiotherapy
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy (N=3)
Abdominal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
Neck edema (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Skin laceration
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Rash on upper extremities
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT04473937/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT04473937/ICF_001.pdf